CLINICAL TRIAL: NCT02670811
Title: Randomized Double-blind Controlled Clinical Study of the Antihypertensive Effect of Fermented Milk With Lactococcus Lactis NRRL-B50571
Brief Title: Antihypertensive Effect of Fermented Milk With Lactococcus Lactis on Prehypertensive Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Investigación en Alimentación y Desarrollo A.C. (Other)
Responsible Party: Principal Investigator, Belinda Vallejo Galland, PhD, PhD, Centro de Investigación en Alimentación y Desarrollo A.C.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VAGB 001
Record Dates: First submitted 2016-01-26; First posted 2016-02-02 (Estimated); Results first posted 2016-10-11 (Estimated); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Hypertension
Keywords: Hypertension; Fermented Milk; Clinical Study; Randomized; Double-blind
MeSH Terms: conditions — Hypertension | interventions — Cultured Milk Products

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Daily consumption of 150 mL of fermented milk with Lactococcus lactis for 8 weeks
  Interventions: Dietary Supplement: Fermented milk
- Placebo (Placebo Comparator): Daily consumption of 150 mL of artificially acidified milk
  Interventions: Dietary Supplement: Acidified milk

INTERVENTIONS:
Dietary Supplement: Fermented milk — 150 mL daily of fermented milk with Lactococcus lactis NRRL-B50571
  Arms: Intervention
Dietary Supplement: Acidified milk — 150 mL daily of artificially acidified milk
  Arms: Placebo

SUMMARY:
The objective of the present work was to evaluate the antihypertensive effect associated with the consumption of fermented milk with Lactococcus lactis NRRL-B50571 on prehypertensive subjects.

DETAILED DESCRIPTION:
A double-blind randomized controlled clinical study of an 8-week intervention with 36 hypertensive subjects was carried out to evaluate the antihypertensive effect of fermented milk with Lactococcus lactis NRRL-B50571. Once obtained the informed consent; volunteers were randomized into two groups (n=18) to either receive 150 mL daily: fermented milk with Lactococcus lactis NRRL-B50571 (intervention group) or artificially acidified milk as control (placebo). Both drinks were consumed daily. Participants were asked not to change their diet or lifestyle during the intervention. We applied intention to treat for those participants who did not have good adherence and those who withdraw the study. The outcomes between groups were analyzed using an independent sample Student t test, with a P value of 0.05 or less (two sided) when there was statistical significance; using statistical software.

ELIGIBILITY:
Inclusion Criteria:

* Systolic blood pressure >130 mmHg
* Diastolic blood pressure > 85 mmHg

Exclusion Criteria:

* Pregnant women
* Cardiovascular diseases
* Diabetes
* Cancer
* Dairy allergy
* Lactose intolerance
* Patients receiving angiotensin converting enzyme inhibitors as pharmacological therapy

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Belinda Vallejo, PhD, Principal Investigator — Centro de Investigación en Alimentación y Desarrollo A.C.

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data for study protocol, statistical analysis plan, clinical study report and analytic code may be shared upon request.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: October 2023 to December 2023.
Access Criteria: Researchers who may benefit for the design on their clinical trial.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who were eligible were asked to sign informed consents. Afterwards all baseline measurements were taken two weeks before randomization and group formations. Subjects who did not fulfill the inclusion criteria were explained why they were not eligible for this study.
Period: Overall Study
Arm/Group | Intervention | Placebo
Started | 18 | 18
Completed | 17 | 18
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Placebo | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.5 (11.7) | 44.6 (9.2) | 42.5 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 10 | 10 | 20
Region of Enrollment [Number; unit: Participants]
  Mexico | 18 | 18 | 36
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 131.8 (5.6) | 134.3 (7) | 133.1 (6.4)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 87.7 (5.1) | 89.3 (5.8) | 88.6 (5.4)
Weight [Mean (Standard Deviation); unit: kilograms] | 80.5 (14.6) | 85.8 (18.2) | 83.2 (16.5)
Height [Mean (Standard Deviation); unit: meters] | 1.63 (0.1) | 1.67 (0.1) | 1.65 (0.1)
Total cholesterol [Mean (Standard Deviation); unit: mg/dL] | 190.1 (43.6) | 178.1 (26) | 184.1 (35.9)
Low density lipoprotein [Mean (Standard Deviation); unit: mg/dL] | 127.1 (43) | 114.7 (26) | 120.9 (35.5)
High density lipoprotein [Mean (Standard Deviation); unit: mg/dL] | 37.9 (8.7) | 37.8 (6.5) | 37.9 (7.6)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] | 137.5 (42.3) | 144.3 (63.5) | 141 (53.3)

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure Measurements
Description: From randomization (baseline), eight weeks of intervention and two weeks after intervention was over.
Time Frame: Baseline to 10 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 18 | 18
mmHg
  Baseline | 131.8 (5.7) | 134.3 (7)
  Week 1 Intake Period | 122.1 (13.6) | 127.4 (11.3)
  Week 2 Intake Period | 121.3 (9.6) | 125.8 (10.3)
  Week 3 Intake Period | 120 (11.4) | 127.1 (8.3)
  Week 4 Intake Period | 121.1 (14.2) | 125 (8.5)
  Week 5 Intake Period | 116.6 (12.3) | 124.8 (11)
  Week 6 Intake Period | 120.4 (11.6) | 126.4 (10.5)
  Week 7 Intake Period | 118.9 (12.6) | 125.6 (10)
  Week 8 Intake Period | 122.5 (8.3) | 127.6 (8.9)
  Week 1 Post-Treatment | 122.3 (12.9) | 127.3 (9.6)
  Week 2 Post-Treatment | 124 (12.6) | 128 (10.2)
Statistical Analysis 1: Comparison: Intervention vs Placebo; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — The primary outcome, systolic blood pressure (mmHg), between groups was analyzed using an independent sample student t test
Statistical Analysis 2: Comparison: Intervention; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — The primary outcome, systolic blood pressure (mmHg), was analyzed using a paired student t test

2. Secondary Outcome: Diastolic Blood Pressure Measurements
Description: From randomization (baseline), eight weeks of intervention and two weeks post-treatment.
Time Frame: Baseline to 10 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 18 | 18
mmHg
  Baseline | 87.7 (5.1) | 89.4 (5.7)
  Week 1 Intake Period | 82.3 (9.5) | 85.9 (7.6)
  Week 2 Intake Period | 80.8 (8) | 84.2 (5.9)
  Week 3 Intake Period | 81.9 (8) | 85.7 (7.9)
  Week 4 Intake Period | 80.4 (10.7) | 84.4 (6.7)
  Week 5 Intake Period | 80.7 (9.1) | 84.5 (8.5)
  Week 6 Intake Period | 82.6 (9.6) | 84.1 (7.8)
  Week 7 Intake Period | 80.7 (11.1) | 84.9 (7)
  Week 8 Intake Period | 83.7 (5.9) | 86.4 (5)
  Week 1 Post-Treatment | 84.3 (9.3) | 87.1 (6.3)
  Week 2 Post-Treatment | 84.7 (9.1) | 86.3 (6.2)
Statistical Analysis 1: Comparison: Intervention vs Placebo; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — The secondary outcome, diastolic blood pressure (mmHg), between groups was analyzed using an independent sample student t test

3. Secondary Outcome: Total Cholesterol Measurements
Description: Total cholesterol in baseline and after 8 weeks of treatment (Intake period).
Time Frame: Baseline and 8th week
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 18 | 18
mg/dL
  Baseline | 190.1 (43.6) | 178.1 (26)
  Week 8 Intake Period | 180.7 (36.1) | 189.8 (39.1)
Statistical Analysis 1: Comparison: Intervention vs Placebo; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — The secondary outcome, total cholesterol (mg/dL), between groups was analyzed using an independent sample student t test

4. Secondary Outcome: Low Density Lipoproteins Measurements
Description: Low density lipoproteins measurements in baseline and after 8 weeks of treatment (intake period).
Time Frame: Baseline and 8th week
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 18 | 18
mg/dL
  Baseline | 127.1 (43) | 114.7 (26)
  Week 8 Intake Period | 116.6 (37.8) | 122.7 (31.8)
Statistical Analysis 1: Comparison: Intervention vs Placebo; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — The secondary outcome, low density lipoprotein (mg/dL), between groups was analyzed using an independent sample student t test

5. Secondary Outcome: High Density Lipoproteins
Description: High density lipoproteins measurements in baseline and after 8 weeks of treatment (intake period).
Time Frame: Baseline and 8th week
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 18 | 18
mg/dL
  Baseline | 37.9 (8.7) | 37.8 (6.5)
  Week 8 Intake Period | 43.2 (8.1) | 42.4 (7.6)
Statistical Analysis 1: Comparison: Intervention vs Placebo; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — The secondary outcome, high density lipoproteins (mg/dL), between groups were analyzed using an independent sample student t test

6. Secondary Outcome: Triglycerides Measurements
Description: Triglycerides measurements in baseline and after 8 weeks of treatment (intake period).
Time Frame: Baseline and 8th week
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 18 | 18
mg/dL
  Baseline | 137.5 (42.3) | 144.3 (63.5)
  Week 8 Intake Period | 103.6 (44.3) | 124.9 (56)
Statistical Analysis 1: Comparison: Intervention vs Placebo; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — The secondary outcome, triglycerides (mg/dL), between groups was analyzed using an independent sample student t test

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Intervention | Placebo
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes